CLINICAL TRIAL: NCT05069129
Title: A Randomized, Controlled Phase I and Sequential Study to Evaluate the Safety and Immunogenicity Following Immunization of GEN2-Recombinant COVID-19 Vaccine (CHO Cells,NVSI-06-08) and Inactivated COVID-19 Vaccine (Vero Cells) in Population Aged 18 Years and Above
Brief Title: Clinical Trial on Sequential Immunization of Recombinant COVID-19 Vaccine (CHO Cells,NVSI-06-08) and Inactivated COVID-19 Vaccine (Vero Cells) in Population Aged 18 Years and Above
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: China National Biotec Group Company Limited (Industry); Lanzhou Institute of Biological Products Co., Ltd (Industry); Beijing Insitute of Biological Products Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CNBG-REC-2021003
Record Dates: First submitted 2021-10-03; First posted 2021-10-06 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Pneumonia; Coronavirus Infections
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subject last vaccination time is within 4-6 months（sequential clinical trial group） (Experimental): Subject have been vaccinated with two doses of Inactivated COVID-19 vaccine (Vero cell).The last vaccination time is within 4-6 months
  Interventions: Biological: Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-08); Biological: Inactivated COVID-19 vaccine (Vero cells)
- Subject last vaccination time is within 7-9 months（sequential clinical trial group） (Experimental): Subject have been vaccinated with two doses of Inactivated COVID-19 vaccine (Vero cell).The last vaccination time is within 91-180 days 7-9 months
  Interventions: Biological: Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-08); Biological: Inactivated COVID-19 vaccine (Vero cells)
- Subject last vaccination time more than 9 months（sequential clinical trial group） (Experimental): Subject have been vaccinated with two doses of Inactivated COVID-19 vaccine (Vero cell).The last vaccination time more than 9 months
  Interventions: Biological: Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-08); Biological: Inactivated COVID-19 vaccine (Vero cells)
- Safety Observation Group (Experimental): Subject have been vaccinated with three doses of Recombinant COVID-19 Vaccine (CHO Cells,NVSI-06-08) on 0，30，60 days
  Interventions: Biological: 3 doses Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-08)

INTERVENTIONS:
Biological: Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-08) — Intramuscular injection of Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-08) in the deltoid muscle of the upper arm
  Arms: Subject last vaccination time is within 4-6 months（sequential clinical trial group）; Subject last vaccination time is within 7-9 months（sequential clinical trial group）; Subject last vaccination time more than 9 months（sequential clinical trial group）
Biological: Inactivated COVID-19 vaccine (Vero cells) — Intramuscular injection of Inactivated COVID-19 vaccine (Vero cells) in the deltoid muscle of the upper arm
  Arms: Subject last vaccination time is within 4-6 months（sequential clinical trial group）; Subject last vaccination time is within 7-9 months（sequential clinical trial group）; Subject last vaccination time more than 9 months（sequential clinical trial group）
Biological: 3 doses Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-08) — Intramuscular injection of Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-08) in the deltoid muscle of the upper arm on 0，30，60 days
  Arms: Safety Observation Group

SUMMARY:
This is randomized, blinded and controlled design. Among the randomly selected subjects who have been vaccinated with two doses of Inactivated COVID-19 vaccine (Vero cell), based on a step-wise approach, the subjects will receive one dose of recombinant COVID-19 vaccine sequentially at different shedules of 4-6 months, 7-9 months and >9 months after two doses of vaccination, and the subjects vaccinated at different schedules will be randomly assigned to different sequential immunization groups. At the same time, each sequential immunization group will be matched with a control group with the inactivated COVID-19 vaccine (vero cells) as the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Age range: populations aged 18 years and above;
* Judged by the investigator that the health condition is well after inquiry and physical examination;
* Vaccinated with 2 doses of CNBG inactivated COVID-19 vaccine according to the product insert（sequential clinical trial group）
* Never vaccinated COVID-19 vaccine（safety observation group）;
* Female subjects who are not nursing or pregnant at the time of enrolment (negative urine pregnancy test) and have no family planning within the first 3 months after enrolment. Effective contraceptive measures have been taken within 2 weeks before inclusion.
* During the whole follow-up period of the study, be able and willing to complete the whole prescribed study plan; Self has ability to understand the study procedures, the informed consent & voluntarily sign an informed consent form and is able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

* Confirmed cases, suspected cases or asymptomatic cases of COVID-19;
* With a history of SARS and MERS infection (self-report, on-site inquiry);
* Has vaccinated with any vaccine other than one or more doses of CNBG inactivated COVID-19 vaccine;
* Axillary temperature ≥ 37.3 ℃ (forehead temperature ≥ 37.8 ℃);
* Previous severe allergic reactions to vaccination (such as acute allergic reactions, urticaria, dyspnea, angioneurotic edema or abdominal pain) or allergy to known components of recombinant COVID-19 vaccine;
* Allergic to any component of the study vaccine (e.g. aluminum, histidine, etc.)
* Known or suspected diseases include：Severe respiratory diseases, severe liver and kidney diseases, hypertension (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 90 mmHg), diabetic complications, malignant tumors, various acute diseases or acute attacks of chronic diseases;
* Has been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* Has a history of convulsions, epilepsy, encephalopathy，long term history of alcohol and drug abuse, history of thyroidectomy, infectious diseasesor mental illness or family history（lineal）;
* With Congenital malformation or developmental disorder, genetic defect, severe malnutrition, etc.;
* Has a history of coagulation dysfunction (e.g. coagulation factors deficiency and coagulation diseases);
* Absence of spleen or splenectomy, functional absence of spleen caused by any condition
* Anti -TB (TB) treatment is under way.
* Patients receiving immunoenhancement or inhibitor therapy within 3 months (continuous oral or IV administration for more than 14 days);
* Received blood products before within 3 months before vaccination;
* Received other investigational drugs within 6 months before vaccination;
* Plan to move before the end of the study or leave the local area for a long time during the scheduled study visit
* Other circumstances judged by investigators that are not suitable for this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1848 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
The incidence and serverity of any adverse reactions | within 30 minutes after vaccination
The incidence and serverity of solicited adverse events | within 30 minutes after vaccination
The incidence and serverity of solicited adverse reactions | within 0-7 days after vaccination
The incidence and severity of unsolicited adverse reactions | within 0-7 days after vaccination
The incidence and serverity of solicited adverse reactions | within 8-30 days after vaccination
The incidence and serverity of solicited adverse events | within 8-30 days after vaccination
The incidence of SAE observed | after vaccination and up to 6 months after full course of immunization.
The incidence of AESI observed | after vaccination and up to 6 months after full course of immunization
GMT of subject's anti- SARS-CoV-2 neutralizing antibody | 15th day after vaccination
GMT of subject's anti- SARS-CoV-2 neutralizing antibody | 30th day after vaccination
Rate of 4-fold rise of anti- SARS-CoV-2 neutralizing antibody | 15th day after vaccination
Rate of 4-fold rise of anti- SARS-CoV-2 neutralizing antibody | 30th day after vaccination

SECONDARY OUTCOMES:
Rate of GMT of subject's anti-SARS-CoV-2 IgG antibody | before vaccination
Rate of GMT of subject's anti-SARS-CoV-2 IgG antibody | 30th day after the full course of vaccination
Rate of 4-fold rise of anti- SARS-CoV-2 neutralizing antibody | before vaccination
Rate of 4-fold rise of anti- SARS-CoV-2 neutralizing antibody | 30th day after the full course of vaccination
GMI of subject's anti-SARS-CoV-2 IgG antibody | before vaccination
GMI of subject's anti-SARS-CoV-2 IgG antibody | 30th day after the full course of vaccination
Proportion of neutralizing antibody titer ≥ 1: 16, ≥ 1: 32 and ≥ 1: 64 | before vaccination
Proportion of neutralizing antibody titer ≥ 1: 16, ≥ 1: 32 and ≥ 1: 64 | 30th day after the full course of vaccination
Rate of Anti-SAR-CoR-2 neutralizing antibody | the 3th month, 6th month, 12th month, 18 month and 24th month after the full course of vaccination
  only sequential clinical trial group
Rate of GMT of IgG antibody | the 3th month, 6th month, 12th month, 18 month and 24th month after the full course of vaccination
  only sequential clinical trial group
Rate of the titer of neutralizing antibody ≥ 1: 16, ≥ 1: 32 and ≥ 1: 64 | the 3th month, 6th month, 12th month, 18 month and 24th month after the full course of vaccination
  only sequential clinical trial group
Rate of Anti-SAR-CoR-2 neutralizing antibody | the 6th month, 12th month after the full course of vaccination
  only Safety Observation Group
Rate of GMT of IgG antibody | the 6th month, 12th month after the full course of vaccination
  only Safety Observation Group
Rate of the titer of neutralizing antibody ≥ 1: 16, ≥ 1: 32 and ≥ 1: 64 | the 6th month, 12th month after the full course of vaccination
  only Safety Observation Group

OTHER OUTCOMES:
The vaccine efficay of recombinant COVID-19 vaccine (CHO cells) against COVID-19, severe cases and deaths | 14th day after vaccination
Anti-SARS-CoV-2 neutralizing antibody | 3th month, 6th month, 9th month and 12th month after full course of immunization
Anti-SARS-CoV-2 GMT of IgG antibody | 3th month, 6th month, 9th month and 12th month after full course of immunization
Proportion of neutralizing antibody titer ≥ 1: 16, ≥ 1: 32 and ≥ 1: 64 | 3th month, 6th month, 9th month and 12th month after full course of immunization
The vaccine efficacy of recombinant COVID-19 vaccine (CHO cells，NVSI-06-08) against COVID-19, severe cases and deaths aged 18 years and above | 15th day after full course of immunization
To evaluate the vaccine efficacy of recombinant COVID-19 vaccine (CHO cells，NVSI-06-08) against different variants after sequential vaccination at different schedules | 15th day after full course of immunization
  only sequential clinical trial group

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Khalifa Medical City, SEHA, Abu Dhab, United Arab Emirates

REFERENCES:
- [Derived] Kaabi NA, Yang YK, Du LF, Xu K, Shao S, Liang Y, Kang Y, Su JG, Zhang J, Yang T, Hussein S, ElDein MS, Yang SS, Lei W, Gao XJ, Jiang Z, Cong X, Tan Y, Wang H, Li M, Mekki HM, Zaher W, Mahmoud S, Zhang X, Qu C, Liu DY, Zhang J, Yang M, Eltantawy I, Hou JW, Lei ZH, Xiao P, Wang ZN, Yin JL, Mao XY, Zhang J, Qu L, Zhang YT, Yang XM, Wu G, Li QM. Safety and immunogenicity of a hybrid-type vaccine booster in BBIBP-CorV recipients in a randomized phase 2 trial. Nat Commun. 2022 Jun 27;13(1):3654. doi: 10.1038/s41467-022-31379-0. PMID 35760812